CLINICAL TRIAL: NCT04659213
Title: Esophagus Deviation During Radiofrequency Ablation of Atrial Fibrillation - EASY AF STUDY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: S4 Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: EASY AF
Record Dates: First submitted 2020-12-02; First posted 2020-12-09 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: This is a prospective, multicenter, randomized controlled, double blinded clinical study to assess a reduction of esophageal lesions attributable to radiofrequency (RF) ablation with use of esolution (esophageal retractor) in comparison to conventional therapy (no use of an esophageal retractor). The randomization is with a 1:1 randomization scheme assigning consecutive patients who meet inclusion and exclusion criteria to either: placement of a luminal esophageal temperature probe(LET) (control group); or, to placement of a LET and insertion of esolution esophageal retractor (intervention group). In the control group, there will not be deviation of the esophagus and in the intervention group, esolution will be utilized to deviate the esophagus during RF catheter ablation. All randomized subjects will be included in the intent-to-treat population, which will be used in the primary study analysis.
Who Masked: Participant, Outcomes Assessor
Masking Description: The study subjects will not know which treatment arm they were randomized to. Additionally, the gastroenterologist performing the endoscopy post-procedure will also be blinded to the treatment arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Interventional Group (Experimental): Placement of a luminal esophageal temperature probe (LET) and insertion of esolution esophageal retractor. In the intervention group, esolution will be utilized to deviate the esophagus during RF catheter ablation
  Interventions: Device: esolution catheter
- Control Group (No Intervention): Placement of a luminal esophageal temperature probe (LET) during RF ablation

INTERVENTIONS:
Device: esolution catheter — esolution is a catheter-based therapy designed to displace the esophagus away from the source of ablation energy during ablation of AF and to eliminate the risk of esophageal injury
  Arms: Interventional Group

SUMMARY:
To assess if deviating the esophagus will reduce/eliminate ablation injury to the esophagus.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age ≥ 22 years and < 80 years
* Clinical decision to proceed with AF ablation procedure.
* Ablation procedure to be completed with General Anesthesia
* Ablation procedure to be completed with use of radiofrequency catheter ablation

Exclusion Criteria:

* History of various esophageal pathology such as esophageal achalasia, varices, strictures, web, carcinoma, tumor/mass, scleroderma, Mallory-Weiss tear, Barrett's esophagitis, diverticulum, banding, laceration, perforation, balloon dilatation.
* Presence of a pH probe deployed in the esophagus
* Planned AF ablation procedure to be completed with laser energy or with cryo-energy
* Acute or uncontrolled psychiatric illness
* Unable to undergo upper endoscopy
* Enrollment in another FDA clinical trial
* Unstable medical condition(s) that precludes safely completing study protocol
* Subject is incarcerated
* Subject is pregnant
* Subject is unable to comprehend the details of the study
* The Investigator believes that the subject will be unwilling or unable to comply with study protocol requirements, including the investigational device procedure and study-related follow up visit requirements

Ages: 22 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Incidence of esophageal injury attributable to RF ablation energy as noted on post ablation endoscopy | 15-72 hours post-ablation procedure
  The primary study endpoint is the incidence of esophageal injury attributable to RF ablation energy as noted on post ablation endoscopy

CONTACTS AND LOCATIONS:
Locations (1):
- OSU, Columbus, Ohio, United States